CLINICAL TRIAL: NCT05037825
Title: The Gut Microbiome and Immune Checkpoint Inhibitor Therapy in Solid Tumors
Acronym: PARADIGM
Status: Recruiting | Type: Observational
Sponsor: VastBiome (Industry)
Responsible Party: Sponsor
Other Study IDs: Pro00054854
Record Dates: First submitted 2021-08-02; First posted 2021-09-08 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Non-Small-Cell Lung Carcinoma; Malignant Melanoma; Renal Cell Carcinoma; Triple-Negative Breast Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Melanoma; Carcinoma, Renal Cell; Triple Negative Breast Neoplasms | interventions — Immune Checkpoint Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Checkpoint Inhibitor, Immune — anti-PD-1, anti-PD-L1, or anti-CTLA-4 as a single agent or in combination with another checkpoint inhibitor or other treatment agent or modality (e.g., targeted therapy, chemotherapy, surgery, radiation, etc.) in accordance with FDA-labeled use of the agent

SUMMARY:
The microbiome has the potential to serve as a robust biomarker of clinical response to immunotherapy. Additionally, microbial manipulation, through diet, exercise, prebiotics, probiotics, or microbially-derived metabolites, may prove to be beneficial in promoting anti-tumor immune responses. However, large prospective studies in humans with longitudinal sample collection and standardized methods are needed to understand how microbiota and their byproducts affect cancer therapies, particularly among patients undergoing identical therapy but experiencing different outcomes. The proposed observational study builds upon these hypotheses by proposing a large cohort design to further assess the associations between the gut microbiota (composition and function), host immune system, and ICI treatment efficacy across multiple cancer types.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women ≥18 years of age
2. Screened negative for COVID-19 symptoms at time of consent, as per institutional policy and as applicable for the duration of the COVID-19 pandemic
3. Diagnosed with stages I-IV primary NSCLC, MM, TNBC or RCC
4. Plan to be treated at a partner cancer site with a checkpoint inhibitor (anti-PD-1, anti-PD-L1, or anti-CTLA-4) as a single agent or in combination with another checkpoint inhibitor or other treatment agent or modality (e.g., targeted therapy, chemotherapy, surgery, radiation, etc.) in accordance with FDA-labeled use of the agent
5. Able to provide informed consent and answer study questionnaires in either English or Spanish
6. Able to provide stool specimens for research purposes

Exclusion Criteria:

1. Mental incapacity
2. Incarcerated individuals
3. Pregnancy (by self-report of pregnancy status)
4. Experiencing active brain metastasis/metastases
5. Treatment with checkpoint inhibitor in off-label capacity or through a clinical/interventional trial
6. Active participation in an immuno-oncology clinical/interventional trial or pharma-sponsored observational study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigator propose to enroll 800 cancer patients (NSCLC, MM, RCC, and TNBC; any stage) who are about to begin standard of care ICI therapy into a multi-site prospective observational study of the gut microbiome.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2021-11-22 (Actual); Primary Completion 2023-09-14 (Estimated); Study Completion 2028-09-14 (Estimated)

PRIMARY OUTCOMES:
Change in microbiome composition from baseline to after Cycle 2 of checkpoint therapy (6-8 weeks) by analyzing longitudinally-collected stool specimens of 800 patients with primary NSCLC, MM, RCC, and TNBC | prior to initiation of checkpoint therapy (i.e. "Baseline") and at the end of Cycle 2 of checkpoint blockade immunotherapy (at approximately 6-8 weeks) ]
  Microbiome evaluation with whole metagenome shotgun sequencing to assess changes in the relative abundance of microbial taxa (measured as percentage abundance per microbial species and changes in percentage abundance between baseline and cycle 2 timepoints) in patients who are receiving checkpoint blockade immunotherapy as the standard of care

SECONDARY OUTCOMES:
Microbiome samples correlation | Time Frame: prior to initiation of checkpoint therapy (i.e. "Baseline") and at the end of Cycle 2 (at approximately 6-8 weeks)
  Definition of a correlation between the gut microbiome and circulating cytokines (specifically IL-2, IL-10, TNF-alpha, IFN-gamma, and G-CSF) and therapeutic response (defined using RECIST criteria).
Microbiome correlation to blood biomarkers | Time Frame: prior to initiation of checkpoint therapy (i.e. "Baseline") and at the end of Cycle 2 (at approximately 6-8 weeks)
  Definition of a correlation between the gut microbiome (measured as percent abundance of microbial taxa derived from whole-metagenome shotgun sequencing) and plasma metabolites (measured in m/z and peak intensities and--where possible--compound abundances in ng/mL) and circulating cytokines (measured in pg/mL per cytokine) in patients receiving checkpoint blockade immunotherapy.
Blood samples correlation | Time Frame: prior to initiation of checkpoint therapy (i.e. "Baseline") and at the end of Cycle 2 (at approximately 6-8 weeks)
  Definition of a correlation between plasma metabolites (measured in m/z and peak intensities and--where possible--compound abundances in ng/mL) and circulating cytokines (measured in pg/mL per cytokine) and therapeutic response (defined using RECIST criteria).

CONTACTS AND LOCATIONS:
Locations (1):
- Baptist Health Clinical Research, Elizabethtown, Kentucky, United States